CLINICAL TRIAL: NCT05010148
Title: Continuous Post-operative Lidocaine Infusion Following Major Reconstructive Spine Surgery in the Elderly to Minimize Delirium and Opiate Use: A Randomized Control Trial
Brief Title: A Clinical Trial of Intravenous Lidocaine After Spinal Surgery to Prevent Delirium and Reduce Pain
Acronym: LIMPP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-32383
Record Dates: First submitted 2021-07-22; First posted 2021-08-18 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Delirium; Postoperative Pain; Spinal Fusion
Keywords: lidocaine; spinal surgery; opioid sparing
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients will be administered D5 water intravenously at the same infusion rate (ml/hr) as the intervention group for 48 hours after major spinal surgery.
  Interventions: Drug: Placebo
- Intervention-Intravenous Lidocaine Infusion (Experimental): Will be administered intravenous lidocaine at 1.33mg/kg/hr (adjusted body weight) for 48 hours following major spinal surgery.
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Lidocaine IV — Intravenous lidocaine will be given at 1.33mg/kg/hr (adjusted body weight) for 48 hours following major spinal surgery
  Other Names: Lidocaine, xylocaine
  Arms: Intervention-Intravenous Lidocaine Infusion
Drug: Placebo — D5 water given at an equivalent ml/hr as intravenous lidocaine (treatment arm) for 48 hours following major spinal surgery
  Other Names: Placebo, D5 water
  Arms: Placebo

SUMMARY:
Postoperative delirium is one of the most frequent adverse events following elective non-cardiac surgery and is associated with cognitive impairment at discharge, as well as in-hospital and long-term mortality, however, despite being a well-recognized problem there is a dearth of effective interventions for prevention and management. A modifiable risk factor associated with postoperative delirium is poor postoperative pain control, and by improving the pain regimen the investigators may be able to decrease the incidence and/or severity of postoperative delirium. In this study, the investigators seek to study whether a postoperative intravenous infusion of lidocaine, known to improve pain control in other contexts, can decrease the risk of postoperative delirium and other opioid-related side effects, following major reconstructive spinal surgery.

DETAILED DESCRIPTION:
Methods:

The investigators will perform a pilot prospective randomized double-blinded placebo-controlled trial of 60 patients undergoing major elective reconstructive spinal surgery to investigate the effect of a postoperative lidocaine infusion on the incidence and severity of postoperative delirium. Major spine surgery is defined as posterior spine fusions >3 levels of instrumentation and fusion, which allows standardization of the level of surgical insult and postoperative analgesic requirements. The intraoperative anesthetic regimen will be standardized to consist of total intravenous anesthesia using sevoflurane, propofol, lidocaine and magnesium (institutional protocol), and fentanyl with boluses allowed per provider discretion.

Patient recruitment, inclusion and exclusion criteria: All surgeons will be contacted before the start of the study to obtain their consent to allow their patients to be studied. The research team has successfully completed multiple National Institutes of Health (NIH) funded cohort and clinical trials at our institution with no surgeon refusing to participate. Eligible patients will be screened from the operating room roster to determine their eligibility. Patients will be contacted by phone or in person for preoperative evaluation. Please see the other section for inclusion and exclusion criteria.

Sample Size Calculation:

The recruitment will be consecutive patients meeting inclusion criteria. Reductions in opioid consumption by ~25% using intravenous lidocaine infusions have been shown to decrease opioid related side effects, but there is essentially no data linking a specific degree of opioid reduction to effects on delirium (46, 47). The most comparable published study to the investigators' proposal is work done by Kaba (2009) studying a lidocaine infusion for abdominal surgery where the average opioid reduction was ~50% (24mg +/-16.3 of piritramide in the placebo vs. 10.33mg +/- 10.33 in the treatment group). Assuming similar reduction in opioids of 50% and similar variance, the proposed sample size, 60 (30 per group), provides a power of 0.8 (alpha = 0.05) to detect a 25% decrease in the use of postoperative opioids.

Randomization: Patients will be randomized utilizing block randomization by a random number generator into either placebo or treatment groups by the research pharmacist. The randomization scheme will be blinded to the researchers and patients.

Anesthetic Management: The anesthetic management will be standardized. All patients will receive a general anesthetic to consisting of 50% oxygen and total intravenous anesthetics consisting of infusions of propofol (60-150 mcg/kg/min), lidocaine (1 mg/kg bolus, then 1.5 mg/kg/hr infusion), magnesium (30 mg/kg bolus, then 6 mg/kg/hr infusion), fentanyl (1 mcg/kg bolus, then 1 mcg/kg/hr infusion, prn boluses), and 0.3 Minimum Alveolar Concentration (MAC) of sevoflurane. Anesthesiologists will be requested to maintain the patient's arterial blood pressure to within 20% of their preoperative baseline using vasoactive agents. Patients will receive mechanical ventilation to maintain normocarbia. Intraoperative warming devices will be used to keep body temperature between 36-37˚C. Oxygen saturation will be maintained >95%. Muscle relaxants will be used during tracheal intubation and only as clinically indicated at other time periods. All patients will be continuously monitored before the induction of anesthesia and during surgery with SEDline Brain Function Monitor (Masimo, Inc., Irvine CA), a standard monitor at our institution. Anesthesiologists will be asked to minimize electroencephalogram (EEG) burst suppression by adjusting the doses of anesthetic drugs since prior studies have suggested a relationship between burst suppression and postoperative delirium (48, 49). Postoperatively, but before discharge from the post anesthetic care unit or upon arrival to the intensive care unit, patients will be randomized to receive either placebo or a lidocaine infusion.

Please see the other sections for a list of primary and secondary outcomes. Briefly the primary outcome is the effect of an intravenous lidocaine infusion on the incidence and severity of postoperative delirium. Secondary outcomes include intravenous lidocaine safety and tolerability, the effect of a lidocaine infusion on opioid usage, pain scores, analgesic satisfaction, opioid related side effects, and functional benefits.

Statistical Analysis The investigators will use descriptive statistics to summarize the characteristics of the study population by treatment groups. The investigators will use an intention to treat paradigm in assessing the effect of the intervention on the outcomes of interest.

Aim 1: To evaluate the safety of a continuous infusion of lidocaine in the first two days after surgery. The investigators will compare the proportion of patients that experienced at least one of the adverse events between the two groups using either the Fisher Exact Test or Chi Square Test as appropriate.

Aim 2: To compare postoperative pain, and opioid usage between patients who receive placebo infusions vs. lidocaine infusions. All opioid doses will be converted to oral morphine equivalents. Specifically, hydromorphone and fentanyl doses will be converted to morphine equivalents using the conversion formula: 1.5 mg of hydromorphone = 10 mg of morphine equivalents, 0.1mg of fentanyl = 10 mg of morphine equivalents (56,57). The investigators will compare the average pain scores and opioids doses between the two treatment groups using two-sample t-tests or Mann-Whitney nonparametric tests if the data are not normally distributed.

Aim 3: To compare the incidence of postoperative delirium between patients who receive placebo infusions vs. lidocaine infusions. Chi-square tests will be conducted to determine the association between lidocaine infusions and incident delirium.

Aim 4: To compare the functional recovery of patients between patients who receive placebo infusions vs. lidocaine infusions. The investigators will compare the results of the 36-Item Short Form Health Survey (SF-36), Oswestry Disability Index (ODI), time to discharge, and ability to participate in physical therapy, using the two sample t-test or Mann-Whitney nonparametric test for continuous outcomes, and Fisher exact Test or Chi Square test for binary outcomes.

Relevant biologic variables - All analyzes will include sex and ethnicity as covariates.

Missing Data - Sensitivity Analyses to Assess the Effects of Missing Data: The investigators will use model-based methods, such as Heckman and Predicted mean matching models to determine the effect of missing observations for each of these reasons on the estimates. The investigators will track the number of missing responses for delirium, and upwardly adjust the sample size accordingly. This strategy may result in having to recruit and follow an additional subject per week in the second year of data collection, which is feasible. The investigators will conduct sensitivity analyses to determine the effect of missing data on the outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

* Elective spinal fusion surgery
* Estimated length of stay ≥3 days
* Fluent in English

Exclusion Criteria:

Surgical:

* Cervical spine surgery
* Non-spine surgeries

Other:

* Allergy or intolerance of lidocaine
* Significant heart disease (2nd or 3rd heart block without a pacemaker, Left ventricular ejection fraction (LVEF) <30%, significant arrhythmia [Adams-strokes, Wolff-Parkinson-white syndrome], concurrent treatment with a class 1 antiarrhythmic or amiodarone)
* Significant hepatic or renal dysfunction
* History of uncontrolled seizures
* Acute porphyria
* Preoperative usage of long-acting opioids (methadone, buprenorphine, fentanyl patch, ms-contin, oxycontin) or preoperative opioid usage greater than or equal to the equivalent of 60 mg of oral morphine equivalents.
* Severe cognitive impairment (reported by proxy or a score of >5 on the Short Portable Mental Status Questionnaire (SPMSQ))
* Self-, or proxy-reported physical impairment preventing the subject from consenting or answering questions
* Evidence of preoperative delirium
* Participated in Clinical Trial of Gabapentin to Decrease Postoperative Delirium and Pain (GIPP) or Postoperative Cognition in Older Adult Surgical Patients (PCD) study previously
* Participating in any other clinical trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Delirium | From 24 hours after start of lidocaine infusion to 3 days after surgery.
  Confusion Assessment Method (CAM) will be performed once daily using a structured interview to assess for delirium incidence. Delirium cases will be validated by a second investigator. Investigators will collect preoperative and surgery related variables that may be associated with delirium.

SECONDARY OUTCOMES:
Severity of Postoperative Delirium | From 24 hours after start of lidocaine infusion to 3 days after surgery.
  To rate delirium severity, the Memorial Delirium Assessment Scale (MDAS) will be used.
Postoperative Opioid Use | From 24 hours after start of lidocaine infusion to discharge, up to one week.
  Postoperative opioids will be measured and abstracted from the electronic medical record. The investigators will convert all opioids to oral morphine equivalents.
Difference in Postoperative Pain Scores Between Treatment Groups | From 8 hours after start of lidocaine infusion to discharge, up to one week.
  Pain will be measured every 8 hours using the 11-point visual analog scale (1=no pain and 10=the worst pain possible) both at rest and with movement preoperatively and daily postoperatively during the hospital admission. In addition, the site and treatment of pain, and the maximal level of pain experienced postoperatively will be measured.
Difference in Analgesic Satisfaction Scores Between Treatment Groups | From 24 hours after start of lidocaine infusion to 3 days after surgery.
  Analgesic satisfaction will be measured daily postoperatively during the hospital admission using the 10-point visual analog scale (1=least satisfied and 10=most satisfied). Patients will be asked daily about the quality of their analgesic regimen and will be asked at their first postoperative follow up appointment with their surgeon.
Difference in Opioid Related Side Effects Between Treatment Groups: Respiratory Depression-Respiratory Rate | From 4 hours after start of lidocaine infusion to discharge, up to one week.
  Respiratory rate will be assessed by reviewing the electronic medical record, with less than 8 breaths per minute defined as respiratory depression.
Difference in Opioid Related Side Effects Between Treatment Groups: Respiratory Depression-Saturated Pulse Oximetry | From 4 hours after start of lidocaine infusion to discharge, up to one week.
  Saturate Pulse Oximetry will be assessed by reviewing the electronic medical record, with a saturation less than 95% defined as respiratory depression.
Difference in Opioid Related Side Effects Between Treatment Groups: Respiratory Depression-Naloxone Administration | From 4 hours after start of lidocaine infusion to discharge, up to one week.
  Naloxone administration will be assessed by reviewing the electronic medical record, and naloxone administration will count as respiratory depression.
Difference in Opioid Related Side Effects Between Treatment Groups: Sedation | From 4 hours after start of lidocaine infusion to discharge, up to one week.
  Sedation will be assessed by the Pasero opioid-induced sedation scale.
Difference in Opioid Related Side Effects Between Treatment Groups: Nausea, Vomiting, Constipation-Investigator Assessments | From 4 hours after start of lidocaine infusion to discharge, up to one week.
  Investigators will conduct daily assessments for symptoms of nausea, vomiting, and constipation.
Difference in Opioid Related Side Effects Between Treatment Groups: Nausea, Vomiting, Constipation-Anti-Emetic Administration | From 4 hours after start of lidocaine infusion to discharge, up to one week.
  Administration of anti-emetics will be assessed by reviewing the electronic medical record.
Difference in Opioid Related Side Effects Between Treatment Groups: Pruritus-Investigator Assessment | From 4 hours after start of lidocaine infusion to discharge, up to one week.
  Investigators will conduct daily assessments for symptoms of pruritus.
Difference in Functional Outcome Between Treatment Groups Using Short Form 36 (SF-36) | Baseline and 3 months.
  Functional recovery from spine surgery will be measured by comparing preoperative and postoperative scores on a variety of questionnaires including the Short-Form 36.
Difference in Functional Outcome Between Treatment Groups Using Oswestry Disability Index (ODI) | Baseline and 3 months.
  Functional recovery from spine surgery will be measured by comparing preoperative and postoperative scores on a variety of questionnaires including the Oswestry Disability Index.
Difference in Time to Discharge Between Treatment Groups | End of hospitalization, at time of discharge, approximately 1 week.
  Functional recovery will be assessed in terms of time to discharge from the hospital.
Difference in Ability to Participate in Physical Therapy Between Treatment Groups | From 24 hours after start of lidocaine infusion to 3 days after surgery.
  Functional recovery will be assessed in terms of the patient's ability to participate with postoperative physical therapy monitored by review of daily physical therapy notes.
Difference in Lidocaine Related Adverse Events Between Treatment Groups | From 4 hours after the start of the lidocaine infusion up to 72 hours.
  The difference in lidocaine treatment related adverse events will be assessed with a screening questionnaire of lidocaine toxicity associated symptoms and compared between treatment groups.
Difference in Cognitive Functioning Between Treatment Groups | From 24 hours after start of lidocaine infusion to 3 days after surgery.
  Cognitive function will be measured using the Mini-Mental State Examination (MMSE).
Cognitive Status | From 24 hours after start of lidocaine infusion to 3 days after surgery.
  Cognitive status will be measured preoperatively using the Telephone Interview of Cognitive Status (TICS) assessment.
Difference in Associative Learning Between Treatment Groups (Cognition) | From 24 hours after start of lidocaine infusion to 3 days after surgery.
  Attention, concentration, and perception will be assessed using the digit symbol substitution test.
Difference in Verbal Fluency Between Treatment Groups (Cognition) | From 24 hours after start of lidocaine infusion to 3 days after surgery.
  Verbal and language skills will be assessed using the timed verbal fluency test.
Word List Learning (Cognition) | From 24 hours after start of lidocaine infusion to 3 days after surgery.
  Cognitive domains of memory and learning will be assessed using the word list learning task.

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Buren, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months following publication.
Access Criteria: To other researchers upon request.

REFERENCES:
- [Derived] Buren MA, Theologis A, Zuraek A, Behrends M, Clark AJ, Leung JM. Lidocaine Infusion for the Management of Postoperative Pain and Delirium (LIMPP): protocol for a randomised control trial. BMJ Open. 2022 Jun 6;12(6):e059416. doi: 10.1136/bmjopen-2021-059416. PMID 35667730

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT05010148/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT05010148/ICF_001.pdf